CLINICAL TRIAL: NCT00524147
Title: Drainage of Tuberculous Pleural Effusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Chi-Li Chung, Department of Internal Medicine, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMU92-AE1-B36
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Tuberculous Pleurisy
Keywords: loculated pleural effusion; pigtail drainage; pleural effusion; pleural thickening; tuberculosis
MeSH Terms: conditions — Tuberculosis, Pleural; Pleural Effusion; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pigtail drainage

SUMMARY:
Tuberculous (TB) pleurisy can cause clinical symptoms and pleural fibrosis with resultant residual pleural thickening (RPT). Therapeutic thoracentesis or initial complete drainage in addition to anti-TB drugs have been tried to rapidly relieve dyspnea caused by effusion and to decrease the occurrence of RPT. However, contradictory results are reported without clear reasons. The researchers' hypothesis is that, in addition to anti-TB medications, early effective evacuation of inflammatory exudates with or without fibrinolytic agents may hasten resolution of pleural effusion, reduce the occurrence of RPT and finally improve long-term functional outcome in patients with TB pleurisy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of tuberculous pleurisy

Exclusion Criteria:

* History of invasive procedures directed into the pleural cavity
* Recent severe trauma, hemorrhage, or stroke; bleeding disorder or anticoagulant therapy
* Use of streptokinase in the previous 2 years
* Lack of clinical symptoms caused by effusions

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-10; Primary Completion 2005-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Chest radiography, daily monitoring of the volume of fluid drained, the time needed for resolution of fever and dyspnea, and total amounts of fluid drained, and the length of chest drainage and hospitalization | baseline, daily after treatment within admission

SECONDARY OUTCOMES:
Chest radiography and pulmonary function testing with spirometry | At discharge and at 2, 4, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Li Chung, MD, Principal Investigator — Department of Internal Medicine, Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chung CL, Chen CH, Yeh CY, Sheu JR, Chang SC. Early effective drainage in the treatment of loculated tuberculous pleurisy. Eur Respir J. 2008 Jun;31(6):1261-7. doi: 10.1183/09031936.00122207. Epub 2008 Jan 23. PMID 18216051